CLINICAL TRIAL: NCT06914427
Title: PET/CT Imaging Study With Simultaneous Dual-nuclide Imaging Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20252098-C-1
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Prostatic Neoplasms; Glioma; PARKINSON DISEASE (Disorder)
MeSH Terms: conditions — Prostatic Neoplasms; Glioma; Parkinson Disease | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- before-after study in the same patient (Experimental): Approximately 35 volunteers are planned to be included in this study. The screened subjects will be scanned with a mononuclide 68Ga/11C probe on the first day, a mononuclide 18F probe on the second day, and a dual-nuclide 68Ga/11C+18F probe on the third day, to validate the isolation effect and quantitative accuracy of dual-nuclide synchrotron imaging technology in humans.
  Interventions: Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/CT — Scanning time: acquisition starts 60±10 minutes after 68Ga/18F probe injection; 10-20 minutes after 11C-MET injection; 60 minutes after 11C-CFT injection; Scanning parameters: whole-body imaging (cranial vault to mid-thigh), routine single-nuclide 3 min/bed; dual-nuclide 5-10 min/bed.

SUMMARY:
This is a study using a parallel control approach and is expected to recruit 35 volunteers, including 8 prostate cancer patients, 8 neuroendocrine tumour patients, 8 glioma patients, 8 Parkinson's syndrome patients, and 3 normal volunteers, to undergo dual-nuclide PET/CT imaging and to validate the isolation effect and quantitative accuracy of simultaneous dual-nuclide imaging in humans.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~75 years old (including boundary values); Gender: male or female; Normal volunteers: males weighing ≥50kg, females weighing ≥45kg, and body mass index [BMI = weight (kg)/height 2 (m2)] within the range of 19.0 ~ 26.0kg/m2 (including borderline values); patients with prostate cancer: patients with pathologically-confirmed biochemical relapsed or primary diagnosed prostate cancer with highly suspected systemic metastases on conventional imaging or PSA levels; patients with neuroendocrine tumour patients: patients with NET (G2-G3) or NEC confirmed by pathology and highly suspected of having more than 3 metastases by conventional imaging; patients with glioma: patients with glioma confirmed by pathology or highly suspected by enhanced MRI and proposed to undergo surgical resection; patients with Parkinson's syndrome: patients with high clinical suspicion of Parkinson's syndrome.

Subjects can fully understand and voluntarily participate in this experiment and sign an informed consent form.

Exclusion Criteria:

* Those who cannot tolerate intravenous drug delivery methods (e.g., history of needle and blood sickness); those with alcohol allergy; and those who, in the opinion of the investigator, are unsuitable to undergo or are unable to complete imaging studies such as PET for specific reasons; Under 18 years of age or ECOG score > 2; Less than 1 month after completion of radiotherapy and less than 2 months after completion of octreotide treatment in patients with neuroendocrine tumours; Women during pregnancy and breastfeeding; Practitioners requiring prolonged exposure to radioactive conditions; Serious diseases of heart, kidney, lung, vascular, nervous and mental systems, immunodeficiency diseases and hepatitis/cirrhosis; Participation in other interventional clinical trials within 1 month prior to screening; Presence of other conditions that, in the opinion of the investigator, make participation in this study unsuitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Signal retention | 1 day from injection of the tracer
  using the 68Ga, 11C, 18F individual imaging images as the gold standard and calculating the retention of the letter lesion area number on the 68Ga/18F and 11C/18F separate images
Clearance | 1 day from injection of the tracer
  calculated by using the 68Ga, 11C and 18F individual imaging images as the gold standard, and calculating the signal clearance of the lesion area on the 18F/68Ga and 18F/11C separate images
SUVmax difference values | 1 day from injection of the tracer
  paired t-test comparing the difference in SUVmax values of lesions on gold standard versus 68Ga/18F and 11C/18F separation images

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine,Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No